CLINICAL TRIAL: NCT00762359
Title: A Study to Investigate the Preventive Effect of AG-1749 Against the Recurrence of Gastric And Duodenal Ulcers During Long-Term Treatment With Low Dose Aspirin.
Brief Title: A Safety and Efficacy Study of Lansoprazole in Preventing Aspirin-Induced Gastric and Duodenal Ulcers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: AG-1749 superior to Gefarnate in ulcer prevention
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG-1749-CCT-351; 070494 (Registry Identifier: JapicCTI); U1111-1113-9929 (Registry Identifier: WHO); R100125 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Stomach Ulcer; Duodenal Ulcer
Keywords: Curling Ulcer; Gastric Ulcer; Aspirin; Acetylsalicylic Acid; Drug Therapy
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer | interventions — Lansoprazole; Gefarnate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lansoprazole 15 mg QD (Experimental)
  Interventions: Drug: Lansoprazole
- Gefarnate 50 mg BID (Active Comparator)
  Interventions: Drug: Gefarnate

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole 15 mg, capsules, orally, once daily and gefarnate placebo-matching capsules, orally, twice daily for up to 12 to 30 months.
  Other Names: AG-1749; PREVACID®; Takepron®
  Arms: Lansoprazole 15 mg QD
Drug: Gefarnate — Gefarnate 50 mg, capsules, orally, twice daily and lansoprazole placebo-matching capsules, orally, once daily for up to 12 to 30 months.
  Arms: Gefarnate 50 mg BID

SUMMARY:
The purpose of this study is to determine whether lansoprazole, once daily (QD), compared to gefarnate, twice daily (BID), is effective in preventing the recurrence of gastric and duodenal ulcers in patients receiving long term treatment with low dosage aspirin.

DETAILED DESCRIPTION:
In Japan, low-dose aspirin is one of the commonly prescribed drugs for inhibiting thrombosis and thrombus formation after angina, myocardial infarction, ischemic cerebrovascular disease, coronary artery by-pass surgery and percutaneous transluminal coronary angioplasty in patients. While low-dose aspirin is effective in these cases, its use sometimes causes gastric and duodenal ulcers which can lead to gastrointestinal bleeding, and in worse cases may lead to death.

The purpose of this study is to assess the efficacy of lansoprazole versus gefarnate in patients with a history of gastric or duodenal ulcers receiving daily low dose aspirin therapy.

ELIGIBILITY:
Inclusion Criteria:

* The patient was on low-dose aspirin treatment on the day when consent was obtained, and requires the long-term continuous treatment even after treatment with the investigational drug is started.
* The patient was confirmed to have a history of gastric ulcer or duodenal ulcer.

Exclusion Criteria:

* Endoscopically confirmed gastric and/or duodenal ulcers on Day 1.
* Endoscopically confirmed active upper gastrointestinal hemorrhage on Day 1.
* Current or past history of aspirin-induced asthma or hypersensitivity to nonsteroidal anti-inflammatory drugs.
* Past or planned surgery affecting gastric acid secretion.
* Clinically significant hepatic or renal disorder.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2007-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Takeda
Locations (65):
- Japan (65):
  - Matsudo-shi, Chiba
  - Yotsukaido-shi, Chiba
  - Imabari, Ehime
  - Matsuyama, Ehime
  - Fukui-shi, Fukui
  - Fukuoka, Fukuoka
  - Onga-gun, Fukuoka
  - Gifu, Gifu
  - Fujioka-shi, Gunma
  - Maebashi, Gunma
  - Higashihiroshima-shi, Hiroshima
  - Hiroshima, Hiroshima
  - Kure-shi, Hiroshima
  - Asahikawa-shi, Hokkaido
  - Hakodate-shi, Hokkaido
  - Sapporo, Hokkaido
  - Nishinomiya-shi, Hyōgo
  - Higashiibaraki-gun, Ibaraki
  - Hitachi-Naka, Ibaraki
  - Inashiki-gun, Ibaraki
  - Namegata-shi, Ibaraki
  - Tsuchiura-shi, Ibaraki
  - Yuuki-shi, Ibaraki
  - Hakusan-shi, Ishikawa-ken
  - Kanazawa, Ishikawa-ken
  - Komatsu-shi, Ishikawa-ken
  - Takamatsu, Kagawa-ken
  - Fujisawa-shi, Kanagawa
  - Kawasaki-shi, Kanagawa
  - Yamato-shi, Kanagawa
  - Yokohama, Kanagawa
  - Yokosuka-shi, Kanagawa
  - Kochi, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Matsusaka-shi, Mie-ken
  - Shima-shi, Mie-ken
  - Tsu, Mie-ken
  - Sendai, Miyagi
  - Ebino-shi, Miyazaki
  - Miyazaki, Miyazaki
  - Jōetsu, Niigata
  - Niigata, Niigata
  - Beppu-shi, Ooita
  - Ōita, Ooita
  - Ibaraki-shi, Osaka
  - Matsubara-shi, Osaka
  - Osaka, Osaka
  - Takatsuki-shi, Osaka
  - Hanyuu-shi, Saitama
  - Ōtsu, Shiga
  - Hamada-shi, Shimane
  - Sunto-gun, Shizuoka
  - Shimotsuke-shi, Tochigi
  - Chiyoda-ku, Tokyo
  - Chuuo-ku, Tokyo
  - Hachioji-shi, Tokyo
  - Kiyose-shi, Tokyo
  - Minato-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Toshima-ku, Tokyo
  - Higashitagawa-gun, Yamagata
  - Iwakuni-shi, Yamaguchi
  - Shimonoseki-shi, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at sites in Japan from May 2007 to November 2008.
Pre-assignment Details: Participants were enrolled in either lansoprazole, once daily (QD) or gefarnate, twice daily (BID) treatment groups.
Groups:
- Lansoprazole 15 mg QD: Lansoprazole 15 mg, capsules, orally, once daily and gefarnate placebo-matching capsules, orally, twice daily for up to 12 to 30 months.
- Gefarnate 50 mg BID: Gefarnate 50 mg, capsules, orally, twice daily and lansoprazole placebo-matching capsules, orally, once daily for up to 12 to 30 months.
Period: Overall Study
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Started | 226 | 235
Completed | 167 | 178
Not Completed | 59 | 57
Not completed — Adverse Event | 20 | 23
Not completed — Protocol Violation | 21 | 13
Not completed — Withdrawal by Subject | 13 | 10
Not completed — Lack of Efficacy | 0 | 4
Not completed — Institution closed | 2 | 3
Not completed — Physician Decision | 2 | 3
Not completed — Removal | 0 | 1
Not completed — Withdrew consent | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID | Total
Number analyzed (Participants) | 226 | 235 | 461
Age, Customized [Number; unit: participants]
  <=39 years | 1 | 0 | 1
  Between 40 and 49 years | 1 | 4 | 5
  Between 50 and 59 years | 31 | 36 | 67
  Between 60 and 64 years | 28 | 32 | 60
  Between 65 and 69 years | 38 | 53 | 91
  Between 70 and 79 years | 105 | 81 | 186
  <=80 years | 22 | 29 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 43 | 94
  Male | 175 | 192 | 367
Region of Enrollment [Number; unit: participants]
  Japan | 226 | 235 | 461

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Gastric Ulcer and/or Duodenal Ulcer
Description: The number of participants that developed gastric ulcer and/or duodenal ulcer at month 18 or final visit. Ulcers are defined as mucosal defect with white coating 3 mm or greater.
Time Frame: 18 Months
Population: Participants not taking investigational drug were not included.
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 226 | 234
participants | 6 | 53
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.0989, 95% CI 2-sided [0.0425 to 0.2300]

2. Secondary Outcome: Change From Baseline in Gastric Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 3)
Description: The Lanza score (partially revised) attributes the severity of induced erosive mucosal injury in the stomach, graded on a 5 point scale (0=normal; 1= erosion/hemorrhage in one area of the stomach and <1 lesion; 2= erosion/hemorrhage in one area of the stomach with 2-5 lesions; 3= erosion/hemorrhage in two areas in the stomach/one area involves >6 lesions; 4= erosion/hemorrhage appear in three or more areas in the stomach). Erosions are mucosal defect < 3 mm. Ulcers are mucosal defect with white coating ≥ 3 mm. Higher scores indicate greater severity of gastric mucosal injury.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 213 | 215
scores on a scale | -0.150 (0.904) | 0.460 (1.241)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change From Baseline in Gastric Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 6)
Description: as for outcome 2
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Median (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 170 | 134
scores on a scale | -0.153 (1.172) | 0.530 (1.444)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change From Baseline in Gastric Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 9)
Description: as for outcome 2
Time Frame: Baseline and Month 9.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 87 | 74
scores on a scale | -0.149 (1.157) | 0.419 (1.375)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0079, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change From Baseline in Gastric Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 12)
Description: as for outcome 2
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 67 | 44
scores on a scale | -0.224 (1.112) | 0.205 (1.047)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0433, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change From Baseline in Gastric Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 18)
Description: as for outcome 2
Time Frame: Baseline and Month 18.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Duodenal Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 3)
Description: The Lanza score (partially revised) attributes the severity of induced erosive mucosal injury in the duodenum, graded on a 4 point scale (0=normal; 1= erosion and hemorrhage are localized in one area of the duodenum and < 1 lesion; 2= 2 to 5 lesions ; 3= > 6 lesions). Erosions are defined as mucosal defect < 3 mm. Ulcers are defined as mucosal defect with white coating ≥ 3 mm. Higher scores indicate greater severity of duodenal mucosal injury.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 212 | 215
scores on a scale | -0.132 (0.552) | 0.228 (0.755)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change From Baseline in Duodenal Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 6)
Description: as for outcome 7
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 170 | 134
scores on a scale | -0.165 (0.583) | 0.149 (0.741)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0006, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change From Baseline in Duodenal Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 9)
Description: as for outcome 7
Time Frame: Baseline and Month 9.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 87 | 74
scores on a scale | -0.092 (0.542) | 0.216 (0.688)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0025, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change From Baseline in Duodenal Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 12)
Description: as for outcome 7
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 67 | 44
scores on a scale | -0.254 (0.766) | 0.136 (0.409)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0010, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change From Baseline in Duodenal Mucosal Injury Assessed by Lanza Score (Partially Revised) (Month 18)
Description: as for outcome 7
Time Frame: Baseline and Month 18.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With Gastric or Duodenal Ulcer or Gastric or Duodenal Hemorrhagic Lesion (Upper Gastrointestinal Hemorrhage)
Description: Number of participants with gastric or duodenal ulcer or gastric or duodenal hemorrhagic lesion (upper gastrointestinal hemorrhage) from baseline through month 18 or final visit. Ulcers are defined as mucosal defect with white coating 3 mm or greater.
Time Frame: 18 Months
Population: Values are from the Full Analysis Set.
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 226 | 234
participants | 7 | 56
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p < 0.0001, Log Rank

13. Secondary Outcome: Change From Baseline in Severity of Postprandial Pain Gastrointestinal Symptom (Month 3)
Description: Postprandial pain is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 202 | 196
scores on a scale | -0.005 (0.187) | 0.015 (0.295)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.6148, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Change From Baseline in Severity of Postprandial Pain Gastrointestinal Symptom (Month 6)
Description: as for outcome 13
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 158 | 133
scores on a scale | -0.025 (0.158) | -0.030 (0.171)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.8050, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Change From Baseline in Severity of Postprandial Pain Gastrointestinal Symptom (Month 9)
Description: as for outcome 13
Time Frame: Baseline and Month 9.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 111 | 86
scores on a scale | -0.027 (0.163) | -0.023 (0.152)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.8678, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Change From Baseline in Severity of Postprandial Pain Gastrointestinal Symptom (Month 12)
Description: as for outcome 13
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 49 | 28
scores on a scale | -0.020 (0.143) | -0.071 (0.262)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.2688, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Change From Baseline in Severity of Postprandial Pain Gastrointestinal Symptom (Month 18)
Description: as for outcome 13
Time Frame: Baseline and Month 18.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 3 | 1
scores on a scale | -0.333 (0.577) | -1.000 (NA) — No test was performed when the number of cases was 5 or less.

18. Secondary Outcome: Change From Baseline in Severity of Hunger and Nighttime Pain Gastrointestinal Symptom (Month 3)
Description: Hunger and nighttime pain is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 202 | 196
scores on a scale | 0.005 (0.307) | 0.026 (0.357)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.7054, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Change From Baseline in Severity of Hunger and Nighttime Pain Gastrointestinal Symptom (Month 6)
Description: as for outcome 18
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 158 | 133
scores on a scale | -0.038 (0.192) | -0.008 (0.261)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.3400, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Change From Baseline in Severity of Hunger and Nighttime Pain Gastrointestinal Symptom (Month 9)
Description: as for outcome 18
Time Frame: Baseline and Month 9.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 111 | 86
scores on a scale | -0.027 (0.211) | -0.023 (0.152)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.8813, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Change From Baseline in Severity of Hunger and Nighttime Pain Gastrointestinal Symptom (Month 12)
Description: as for outcome 18
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 49 | 28
scores on a scale | 0.000 (0.204) | -0.071 (0.262)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.1862, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Change From Baseline in Severity of Hunger and Nighttime Pain Gastrointestinal Symptom (Month 18)
Description: as for outcome 18
Time Frame: Baseline and Month 18.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 3 | 1
scores on a scale | -0.333 (0.577) | -1.000 (NA) — No test was performed when the number of cases was 5 or less.

23. Secondary Outcome: Change From Baseline in Severity of Feeling of Enlarged Abdomen Gastrointestinal Symptom (Month 3)
Description: Feeling of enlarged abdomen is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 202 | 196
scores on a scale | -0.020 (0.315) | -0.005 (0.312)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.8604, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Change From Baseline in Severity of Feeling of Enlarged Abdomen Gastrointestinal Symptom (Month 6)
Description: as for outcome 23
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 158 | 133
scores on a scale | -0.019 (0.329) | 0.015 (0.325)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.5485, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: Change From Baseline in Severity of Feeling of Enlarged Abdomen Gastrointestinal Symptom (Month 9)
Description: as for outcome 23
Time Frame: Baseline and Month 9.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 111 | 86
scores on a scale | -0.027 (0.368) | -0.023 (0.265)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.7382, Wilcoxon (Mann-Whitney)

26. Secondary Outcome: Change From Baseline in Severity of Feeling of Enlarged Abdomen Gastrointestinal Symptom (Month 12)
Description: as for outcome 23
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 49 | 28
scores on a scale | -0.020 (0.143) | -0.036 (0.331)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.7619, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Change From Baseline in Severity of Feeling of Enlarged Abdomen Gastrointestinal Symptom (Month 18)
Description: as for outcome 23
Time Frame: Baseline and Month 18.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 3 | 1
scores on a scale | NA (NA) — No test was performed when the number of cases was 5 or less. | NA (NA) — No test was performed when the number of cases was 5 or less.

28. Secondary Outcome: Change From Baseline in Severity of Feeling of Nausea Gastrointestinal Symptom (Month 3)
Description: Feeling of nausea is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 202 | 196
scores on a scale | -0.025 (0.233) | 0.020 (0.142)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0204, Wilcoxon (Mann-Whitney)

29. Secondary Outcome: Change From Baseline in Severity of Feeling of Nausea Gastrointestinal Symptom (Month 6)
Description: as for outcome 28
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 158 | 133
scores on a scale | -0.051 (0.220) | 0.008 (0.087)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0046, Wilcoxon (Mann-Whitney)

30. Secondary Outcome: Change From Baseline in Severity of Feeling of Nausea Gastrointestinal Symptom (Month 9)
Description: as for outcome 28
Time Frame: Baseline and Month 9.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 111 | 86
scores on a scale | -0.072 (0.260) | 0.012 (0.108)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0059, Wilcoxon (Mann-Whitney)

31. Secondary Outcome: Change From Baseline in Severity of Feeling of Nausea Gastrointestinal Symptom (Month 12)
Description: as for outcome 28
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 49 | 28
scores on a scale | -0.082 (0.277) | 0.000 (0.000)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.1229, Wilcoxon (Mann-Whitney)

32. Secondary Outcome: Change From Baseline in Severity of Feeling of Nausea Gastrointestinal Symptom (Month 18)
Description: as for outcome 28
Time Frame: Baseline and Month 18.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 3 | 1
scores on a scale | NA (NA) — No test was performed when the number of cases was 5 or less. | NA (NA) — No test was performed when the number of cases was 5 or less.

33. Secondary Outcome: Change From Baseline in Severity of Feeling of Heartburn Gastrointestinal Symptom (Month 3)
Description: Feeling of heartburn is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 202 | 196
scores on a scale | -0.064 (0.387) | -0.005 (0.411)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.2694, Wilcoxon (Mann-Whitney)

34. Secondary Outcome: Change From Baseline in Severity of Feeling of Heartburn Gastrointestinal Symptom (Month 6)
Description: as for outcome 33
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 158 | 133
scores on a scale | -0.089 (0.346) | 0.038 (0.451)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.0141, Wilcoxon (Mann-Whitney)

35. Secondary Outcome: Change From Baseline in Severity of Feeling of Heartburn Gastrointestinal Symptom (Month 9)
Description: as for outcome 33
Time Frame: Baseline and Month 9.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 111 | 86
scores on a scale | -0.063 (0.411) | 0.000 (0.376)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.3128, Wilcoxon (Mann-Whitney)

36. Secondary Outcome: Change From Baseline in Severity of Feeling of Heartburn Gastrointestinal Symptom (Month 12)
Description: as for outcome 33
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 49 | 28
scores on a scale | -0.163 (0.373) | -0.036 (0.331)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.1450, Wilcoxon (Mann-Whitney)

37. Secondary Outcome: Change From Baseline in Severity of Feeling of Heartburn Gastrointestinal Symptom (Month 18)
Description: as for outcome 33
Time Frame: Baseline and Month 18.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 3 | 1
scores on a scale | NA (NA) — No test was performed when the number of cases was 5 or less. | NA (NA) — No test was performed when the number of cases was 5 or less.

38. Secondary Outcome: Change From Baseline in Severity of Anorexia Gastrointestinal Symptom (Month 3)
Description: Severity of anorexia is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 202 | 196
scores on a scale | 0.005 (0.254) | 0.010 (0.175)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.6175, Wilcoxon (Mann-Whitney)

39. Secondary Outcome: Change From Baseline in Severity of Anorexia Gastrointestinal Symptom (Month 6)
Description: as for outcome 38
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 158 | 133
scores on a scale | -0.019 (0.177) | 0.000 (0.246)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.4496, Wilcoxon (Mann-Whitney)

40. Secondary Outcome: Change From Baseline in Severity of Anorexia Gastrointestinal Symptom (Month 9)
Description: as for outcome 38
Time Frame: Baseline and Month 9.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 111 | 86
scores on a scale | -0.018 (0.190) | 0.000 (0.153)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.4718, Wilcoxon (Mann-Whitney)

41. Secondary Outcome: Change From Baseline in Severity of Anorexia Gastrointestinal Symptom (Month 12)
Description: as for outcome 38
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 49 | 28
scores on a scale | 0.000 (0.204) | -0.036 (0.189)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.4484, Wilcoxon (Mann-Whitney)

42. Secondary Outcome: Change From Baseline in Severity of Anorexia Gastrointestinal Symptom (Month 18)
Description: as for outcome 38
Time Frame: Baseline and Month 18.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 3 | 1
scores on a scale | -0.333 (0.577) | NA (NA) — No test was performed when the number of cases was 5 or less.

43. Secondary Outcome: Change From Baseline in Severity of Hematemesis and Melena Gastrointestinal Symptom (Month 3)
Description: Severity of hematemesis and melena (blood stool, black stool, tarry stool) is graded on a 4 point scale (0=none; 1=mild; 2=moderate; 3=severe). Higher scores indicate greater severity of gastrointestinal symptom.
Time Frame: Baseline and Month 3.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 202 | 196
scores on a scale | -0.010 (0.099) | 0.020 (0.286)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.2604, Wilcoxon (Mann-Whitney)

44. Secondary Outcome: Change From Baseline in Severity of Hematemesis and Melena Gastrointestinal Symptom (Month 6)
Description: as for outcome 43
Time Frame: Baseline and Month 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 158 | 133
scores on a scale | -0.006 (0.138) | 0.000 (0.123)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.6818, Wilcoxon (Mann-Whitney)

45. Secondary Outcome: Change From Baseline in Severity of Hematemesis and Melena Gastrointestinal Symptom (Month 9)
Description: as for outcome 43
Time Frame: Baseline and Month 9.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 111 | 86
scores on a scale | -0.009 (0.165) | -0.012 (0.108)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.9015, Wilcoxon (Mann-Whitney)

46. Secondary Outcome: Change From Baseline in Severity of Hematemesis and Melena Gastrointestinal Symptom (Month 12)
Description: as for outcome 43
Time Frame: Baseline and Month 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 49 | 28
scores on a scale | -0.020 (0.143) | 0.000 (0.000)
Statistical Analysis 1: Comparison: Lansoprazole 15 mg QD vs Gefarnate 50 mg BID; Test type: Superiority or Other; p = 0.4497, Wilcoxon (Mann-Whitney)

47. Secondary Outcome: Change From Baseline in Severity of Hematemesis and Melena Gastrointestinal Symptom (Month 18)
Description: as for outcome 43
Time Frame: Baseline and Month 18.
Population: No test was performed when the number of cases was 5 or less. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 3 | 1
scores on a scale | NA (NA) — No test was performed when the number of cases was 5 or less. | NA (NA) — No test was performed when the number of cases was 5 or less.

48. Secondary Outcome: Number of Participants With Adverse Events
Description: Treatment-emergent adverse events (TEAE) are adverse events with an onset that occurs after receiving study drug. A TEAE may also be a concurrent medical condition diagnosed prior to the date of first dose of study drug that increases in severity after the start of dosing. Please see Other Adverse Events table below for TEAE listings.
Time Frame: 18 Months
Measure: Number; unit: participants
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Number analyzed (Participants) | 226 | 234
participants
  Adverse event | 166 | 168
  Adverse event (Frequency ≥5%) | 82 | 68
  Adverse event related to the study drug | 26 | 25
  Serious adverse event | 27 | 26
  Serious adverse event related to the study drug | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were summarized by onset date occurring on or after the first dose of double-blind study medication.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Lansoprazole 15 mg QD | Gefarnate 50 mg BID
Serious Adverse Events (participants affected / at risk) | 27/226 | 26/234
Other Adverse Events (participants affected / at risk) | 82/226 | 68/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lansoprazole 15 mg QD (N=226) | Gefarnate 50 mg BID (N=234)
Colonic polyp (Gastrointestinal disorders) | 1 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Corneal degeneration (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Angina pectoris (Cardiac disorders) | 4 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Cyst (General disorders) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lansoprazole 15 mg QD (N=226) | Gefarnate 50 mg BID (N=234)
Constipation (Gastrointestinal disorders) | 14 | 8
Diarrhoea (Gastrointestinal disorders) | 19 | 2
Reflux oesophagitis (Gastrointestinal disorders) | 3 | 16
Nasopharyngitis (Infections and infestations) | 51 | 45
Fall (Injury, poisoning and procedural complications) | 13 | 9

LIMITATIONS AND CAVEATS:
On September 2008, the Efficacy and Safety Evaluation Committee recommended that this study be discontinued based on the interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial contract states that information should never be disclosed without prior consent of the sponsor, although it does not specify the number of days during which disclosure of information is limited.